CLINICAL TRIAL: NCT01403363
Title: Use of Fentanyl Patch in Partial Doses Than the Original
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MMC1111311KCTIL
Record Dates: First submitted 2011-07-25; First posted 2011-07-27 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- fentanyl patch (Experimental)
  Interventions: Drug: use of fentanyl patch that was halved

INTERVENTIONS:
Drug: use of fentanyl patch that was halved — A sample of 95 patients will be recruited. Once consent form is signed, blood samples will be collected twice: 1. At the time of the visit; 2. After 144 hours (about 6 days) from the first sample, and at least 36 hours after replacing the cut patch. Pain management will be evaluated at both visits using the Brief Pain Inventory (Hebrew version) - BPI questionnaire, and rescue doses used before and after the cutting of the patch. The blood samples will be transferred to the laboratory for testing of fentanyl concentration levels.

SUMMARY:
Fentanyl is considered a potent synthetic opioid widely used in anesthesiology, for short and long-term pain management, and for sedation. The fentanyl patch is constructed like a matrix, a system based on a polyacrylate net with fentanyl that attaches directly onto the skin. The doses available today are from 12µg/h, 25, 50, 75, to 100 µg/h. Despite the variable doses available, often in certain patients as the elderly or children, there is a need for slower titration than the 12 µg/h currently available.

In this study, the investigators aim to evaluate pain control and to examine the blood fentanyl concentration of patients on a fix dose of fentanyl patch up to 100 µg/h every two or three days, and compare it with pain control and concentration levels obtained from a similar dose patch, but after cutting the patch into two.

The study will take place at the pain clinic of Clalit Health Services-South District (CHS-SD), and the Negev home palliative care unit. In CHS-SD there are approximately 300 patients treated regularly with opioids and about 120 patients in the home palliative care unit. A sample of 95 patients will be recruited. Once consent form is signed, blood samples will be collected twice: 1. At the time of the visit; 2. After 144 hours (about 6 days) from the first sample, and at least 36 hours after replacing the cut patch. Pain management will be evaluated at both visits using the Brief Pain Inventory (Hebrew version) - BPI questionnaire, and rescue doses used before and after the cutting of the patch. The blood samples will be transferred to the laboratory for testing of fentanyl concentration levels.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from chronic pain on a fixed dose of fentanyl patch for over two weeks, with a maximum dose of 100 µg/h every two or three days, and have given their informed consent will be included in the study.

Exclusion Criteria:

* Patients with cognitive problems
* non-Hebrew speaking
* patients that their medical condition prevents them from participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2012-03; Primary Completion 2016-03 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
change of blood concentration levels of fentanyl and nurofentanyl | 1. At the time of the visit; 2. After 144 hours (about 6 days) from the first sample, and at least 36 hours after replacing the cut patch
  2 ml blood samples will be transferred under refrigerated conditions to the lab for a chromatography test using spectrometry testing for fentanyl and nurofentanyl. The change of blood concentration levels of fentanyl and nurofentanyl will be examined.

SECONDARY OUTCOMES:
Change of patients pain assessment | 1. At the time of the visit; 2. After 144 hours (about 6 days) from the first sample, and at least 36 hours after replacing the cut patch
  Pain management will be evaluated at both visits using the Brief Pain Inventory (Hebrew version) - BPI questionnaire. We will examine the change of patients pain assessment

CONTACTS AND LOCATIONS:
Overall Officials: Pesach Shvartzman, MD, Principal Investigator — Clalit Health Services
Locations (1):
- Pain clinic of Clalit Health Services-South District (CHS-SD), Beersheba, Israel